CLINICAL TRIAL: NCT02174809
Title: Curbing Gestational Weight Gain in Primary Care: Using Technology Based on Behaviour Change Theory
Brief Title: Gestational Weight Gain in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helena Piccinini (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Helena Piccinini, Family Physician, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P12PiccVall
Record Dates: First submitted 2014-03-28; First posted 2014-06-26 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Gestational Weight Gain
Keywords: Pregnancy; Gestational Weight Gain; Primary Care; Guidelines
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5As (Experimental): Physicians' use of the 5As tool to discuss gestational weight gain with their pregnant patients
  Interventions: Behavioral: Use of 5As to discuss gestational weight gain
- Usual care (Active Comparator): Usual care by physicians in addressing gestational weight gain with their pregnant patients
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Use of 5As to discuss gestational weight gain
  Other Names: 5As of Healthy Pregnancy Weight Gain
  Arms: 5As
Behavioral: Usual care
  Other Names: Usual care by physicians in addressing gestational weight gain
  Arms: Usual care

SUMMARY:
Excess weight gain in pregnancy is linked to a number of adverse outcomes for mothers and their offspring, and in 2011, 59 % of women in Nova Scotia gained weight in excess of recommendations. A number of factors influence how much weight a woman gains, including lack of knowledge, age, the number of previous pregnancies she's had, smoking, ethnicity, income, and education. Although a clinician's advice also plays a role, simply giving advice does not necessarily translate into patient behaviour change. On the other hand, advice that is given through a patient-centred approach is significantly associated with increased patient acceptance of and adherence to recommendations, and increased intentions and attempts at behaviour change. In addition, this approach has been shown to decrease costs to the health care system. Patient-centredness can measured from the perspective of the clinician, an observer, or the patient. Research suggests that the patient's perspective of patient-centredness is the perspective most significantly associated with improved health outcomes.

Clinicians avoid discussing weight-related matters for a number of reasons, including a lack of time and general discomfort in raising the subject. There are some tools that can address some of these barriers, and example being the "5As of Obesity Management". This tool is based on principles of behaviour change science and patient-centredness. Pilot data on the use of this tool showed a two-fold increase in the initiation of weight-related discussions between clinicians and their patients. Our team was instrumental in the development, dissemination and initial evaluation of this tool, and Dr. Piccinini-Vallis has recently led a national multidisciplinary endeavor to adapt it to pregnancy, which has resulted in the "5As of Healthy Pregnancy Weight Gain" tool. It is now time to evaluate whether the use of this tool is acceptable to clinicians and whether its use translates into any patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Family physicians providing prenatal care
* Patients who are pregnant

Exclusion Criteria:

* Multiple pregnancy
* Abnormal pregnancy
* Inability to read and inability to speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Guideline-concordance of women's total gestational weight gain | 12 months
  The congruence of total gestational weight gain with Institute of Medicine guidelines based on pre-pregnancy body mass index

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Halifax Regional Municipality, Halifax, Nova Scotia
  - Nova Scotia Health Authority, Halifax, Nova Scotia